CLINICAL TRIAL: NCT06323759
Title: Perinatal EDucation: Pedagogical Strategy and Facilitators for the PROMotion of BreastFeeding
Acronym: PED-PROM-BF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lépine Alexandra (Other)
Responsible Party: Sponsor-Investigator, Lépine Alexandra, responsable-bred@univ-paris.fr, Université Sorbonne Paris Nord
Organization: Université Sorbonne Paris Nord (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2022-14
Record Dates: First submitted 2024-03-10; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Breast Feeding
Keywords: Breast Feeding Promotion; Pedagogical Strategy
MeSH Terms: conditions — Breast Feeding | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: This intervention is based on a pedagogical engineering that proposes a favorable learning environment more adapted than the courses already offered in preparing for parenthood and promoting breastfeeding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (No Intervention): Pregnant women have taken a routine parenthood preparation courses and follow-up by independent midwives in antenatally
- INTERVENTION GROUP (Other): Pregnant women have taken a new parenthood preparation courses and follow-up by independent midwives in antenatality, postnatality short term, and postnatality long term)
  Interventions: Other: educational intervention

INTERVENTIONS:
Other: educational intervention — In antenatal breastfeeding education: Theoretical contributions on BF (physiology of lactation, frequency complications), hands-on workshop, Provision of educational tools to promote the learning environment: breastfeeding booklet, educational video on breastfeeding, link to a BF specific platform, access to a telephone platform. In short-term postnatal breastfeeding education: Three systematic fallow-up at home or at midwives' office are planned. During these visits, a time of systematic discussion is planned with the nursing mothers. Their knowledge and ability to manage their breastfeeding are checked. The physiology of lactation, the gestures of breastfeeding and the occurrence of common complications are systematically recalled by the liberal midwife. In long-term postnatal breastfeeding education: Invitation of nursing mothers to breastfeeding information meetings at 2nd and 4th month after birth. These meetings will be facilitated either by the liberal midwives.
  Arms: INTERVENTION GROUP

SUMMARY:
Breastfeeding up to 6 months of a child's life, for its benefits to mother and child, has become a global public health goal. However, there is a disparity in the prevalence of breastfeeding (BF) in different regions of the world. According to French perinatal surveys, the rate of BF at birth decreased significantly between 2010 and 2016. Even if that figure remains stable according to the last perinatal survey in 2021, it decreases sharply, to 34.4%, at 2 months.While many plans at the national level advocate for BF, it is rare to see an action plan or an education intervention for women and couples aimed at promoting BF. However, women's needs to educate about BF and the need for professionals to reflect on their practices are highlighted by numerous perinatal surveys. It should be noted that despite the importance given to the promotion of BF found in all National Nutrition and Health Programs, none of them provide pedagogical means or an education program to achieve the objectives set. At present, in France, there is no breastfeeding education program and professionals accompany women by implementing experimental actions without considering the complexity of the promotional dimension (producing a behavioral change) and the educational dimension (understanding the pedagogy of the proposed actions)

DETAILED DESCRIPTION:
The benefits of exclusive breastfeeding for infants and mothers are widely recognized by the scientific community.

As a result, its promotion has become a global public health goal: 75% of newborns should be breastfed by 2030. According to the World Health Organization (WHO), the global average for exclusive breastfeeding has increased from 14% in 1985 to 37% in 2015. The WHO report also notes a disparity in the prevalence of exclusive breastfeeding at birth and at six months of age.

According to the National Health Nutrition Programs and the recommendations of Public Health France and the French Society of Pediatrics, the promotion of exclusive breastfeeding remains the main preventive measure to combat health inequalities from childhood to ensure healthy and equitable development. They emphasize the education of mothers and/or couples, providing women with "know-how to act" by acquiring knowledge, developing management skills, and building self-confidence and motivation. However, these plans set quantified objectives, but do not propose educational actions or interventions to promote BF, and even less indicate the means for professionals to achieve these objectives.

In France, couples and/or women can, if they wish, benefit from birth and parenting preparation sessions offered by midwives in the prenatal period. One of these sessions is dedicated to encouraging and educating pregnant women to breastfeed. In the postnatal period, despite an increase in the number of staff trained to support breastfeeding mothers, more than 84% of couples are referred to breastfeeding support networks outside the maternity unit (PMI, private midwives, associations). Even the practice of early discharge (stay < 2 days) for low-risk women has inevitably reduced the time spent by hospital staff in educating women. At present, this activity is outsourced and carried out by private midwives, who carry out between 2 and 3 early postnatal follow-up consultations to assess the mother's and newborn's needs on a medical, psycho-educational level. These consultations are not mandatory but are strongly recommended.

Further scientific research:

A scoping review of international publications carried out in 2020 made it possible to draw a map of the pedagogical methods practiced, to identify some of their characteristics favoring the initiation and duration of BF, and to demonstrate that professionals rarely refer to a pedagogical strategy and conditions favorable to learning to ensure a better promotion of BF. The areas for improvement identified can be considered in order to better adapt educational strategies in terms of their pedagogical design. In addition to this literature review, a multicenter and prospective survey will be carried out among breastfeeding women and hospital midwives who led the childbirth preparation sessions to identify, on the one hand, the educational needs of breastfeeding women and, on the other hand, the educational strategies proposed by caregivers to promote BF. This study has been approved by the Ethics Committee of the Sorbonne University N°CER-2021-119 and is registered in the ClinicalTrials.gov registry: NCT05271812.

The survey highlights that, overall, the educational needs expressed by breastfeeding women and the educational approaches taken by midwives correlate with the educational characteristics identified in the Scope Review. Midwives' pedagogical attitudes as well as the educational strategies they propose seem to have an impact on the reinforcement of the decision to breastfeed and the continuation of this decision in the longer term. The perceived usefulness of the educational session is expressed in the reinforcement of the motivation to breastfeed, the development of self-esteem and the feeling of self-management (competence to manage their breastfeeding). We also identified the pedagogical characteristics of the educational sessions offered by midwives. Thus, this review of the literature, coupled with the survey of women's educational strategies and needs, has allowed us to draw up pedagogical guidelines that can be built around a more adapted engineering to promote BF.

Based on the results of the scoping review and the primary study, we modeled an educational intervention based on a strategy, including favorable conditions, to promote breastfeeding.

The research question is therefore: Can an adapted educational intervention based on an educational strategy and conducive learning conditions improve the promotion of breastfeeding? Theoretical framework: This research focuses on the pedagogical dimension and, more specifically, on improving the pedagogical engineering of current educational interventions (in the context of antenatal and postnatal follow-up of women) and their contribution to the maintenance of breastfeeding from the point of view of women and professionals.

This is a systemic approach based on evaluations of therapeutic education programs. It allows for a more comprehensive and different approach to biomedical and clinical research that attempts to demonstrate the effectiveness of a program or intervention in BF promoting without explaining the didactics of the programs.

The evaluation framework of this model is based on critical realism. It is proposed by Greenhalgh, Harvey and Walshe and explained in the RAMESES II reporting standards for realist evaluations. Numerous publications, by Ridde.V and Robert.E, confirm the relevance of the pragmatic approach, which allows researchers to explain what works in a program, for what reasons and in what contexts. It makes it possible to establish an explanatory theory for a program model, according to the contexts that influence it and the mechanisms that hinder effects. Bearing in mind that these operations are not linear and that the expected effects (results) may be different depending on the conditions of time, place, individuals themselves, social, cultural, political, and economic organizations. It is a multi-center, comparative, mixed-methods study with a comprehensive approach. Realistic evaluation shows what works and what does not work in a program, and how and to what effect. It enables the construction of an explanatory theory in terms of contexts of influence, generative mechanisms, and effects produced in the BF ecosystem.

This is a sequential and explanatory mixed-methods study (QUANTI-Quali). Quantitative data will be analyzed using R software, while qualitative data analysis will be conducted using Atlas-Ti software.

ELIGIBILITY:
Inclusion Criteria:

for women for all pregnant women in Control Group & Intervention Group:

* Aged ≥ 18, French-speaking, with access to and use of the internet
* Pregnant woman followed in one of the maternity wards, presenting with a simple pregnancy, physiological course
* Consenting to participate in the research For Liberal Midwives
* Participation on a voluntary basis
* Experience teaching parenting and breastfeeding classes

Exclusion Criteria:

for women for all pregnant women in Control Group & Intervention Group

* Medical-gynecological history requiring medication management incompatible with lactation
* History of breast surgery that contraindicates breastfeeding
* Women without access to the Internet and who do not speak French.
* Women refusing to participate in research.

For Liberal Midwives

- Liberal midwives refusing to participate in research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
To find out the contribution of educational engineering to the choice and continuation of breastfeeding from the point of view of women until 4 months after the birth of the child. | T1: Prenatal: during the 9th month of pregnancy T2: Postnatal: during the 1st week after returning home T3: Postnatal: during the 3rd week of returning home T4: Postnatal: during the 8th week of return home, i.e. 2nd month after the birth of the child
  The percentage of women who are exclusively breastfeeding. They will be asked about their breastfeeding status at 15 days, 1 month, 2 months, and 4 months.

SECONDARY OUTCOMES:
To explain contexts and generative mechanisms of pedagogical design that influence breastfeeding management up to 4 months afther birth. | T2: Postnatal: during the 1st week after returning home T3: Postnatal: during the 3rd week of returning home T4: Postnatal: during the 8th week of return home, i.e. 2nd month after the birth of the child
  To measure women's perception of usefulness in the pedagogical design of the educational intervention for the management of breastfeeding and its complications.Women will be surveyed using closed-ended questions to assess their level of competence in breastfeeding management based on what they have learned, the content of the course, and practice of the gestures they have learned.
  Level of understanding, level of importance felt by breastfeeding women, and level of satisfaction with the courses are measured on a 4-point Likert scale. The level of influence of the courses on women's motivation to continue breastfeeding is measured on a 10-point nuance scale. Closed-ended questions about self-efficacy in breastfeeding management are administered to women.
To explain interactions between existing contexts, generative mechanisms and effects on women's breastfeeding management skills. | T2: Postnatal: during the 1st week after returning home T3: Postnatal: during the 3rd week of returning home T4: Postnatal: during the 8th week of return home, i.e. 2nd month after the birth of the child
  To measure the development of women's conative skills through the educational intervention and in different breastfeeding situations.Women will be interviewed using closed-ended questions to assess their feelings of self-esteem and commitment to breastfeeding based on 9 and 11 items respectively using 10-point nuanced scales. Two open-ended questions about self-esteem and breastfeeding commitment are included so that interviewed women can explain their responses.
To determine contexts and generative mechanisms of pedagogical design that influence women's knowledge of breastfeeding up to 4 months afther birth. | T2: Postnatal: during the 1st week after returning home T3: Postnatal: during the 3rd week of returning home T4: Postnatal: during the 8th week of return home, i.e. 2nd month after the birth of the child
  The perception of learning to manage breastfeeding and its most common complications. Women will be interviewed using closed-ended questions to assess their self-efficacy in managing their breastfeeding. This involves the short version of the breastfeeding self-efficacy scale. Fourteen items are evaluated on a 4-point Likert scale. An open-ended question is included so that interviewed women can explain their responses.

OTHER OUTCOMES:
To evaluate the level of satisfaction about the educational intervention among nursing mothers. | T1: Prenatal: during the 9th month of pregnancy T2: Postnatal: during the 1st week after returning home T3: Postnatal: during the 3rd week of returning home T4: Postnatal: during the 8th week of return home, i.e. 2nd month after the birth of the child
  To evaluate breastfeeding mothers' satisfaction with educational intervention.Women will be interviewed using closed-ended questions to evaluate their satisfaction with the educational intervention for managing their breastfeeding. Women's satisfaction will be assessed using a 4-point Likert scale. An open-ended question is planned so that interviewed women can explain their responses.

CONTACTS AND LOCATIONS:
Overall Officials: Mehrnoosh Yazdanbakhsh, Principal Investigator — Université Sorbonne Paris Nord Laboratoire d'Educations et Promotion de la santé - UR3412; Rémi Gaganyre, Study Director — Université Sorbonne Paris Nord Laboratoire d'Educations et Promotion de la santé - UR3412
Locations (1):
- Université Sorbonne Paris Nord - Laboratoire d'Educations et Promotion de la Santé - UR 3412, Bobigny, France

IPD SHARING:
Plan to Share IPD: No
No individual data collected will be shared with other researchers.